CLINICAL TRIAL: NCT00964353
Title: The Hospital and Economics CERT: Project 1: The Clinical and Economic Implications of Genetic Testing for Warfarin Management
Brief Title: Clinical and Economic Implications of Genetic Testing for Warfarin Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16738B
Record Dates: First submitted 2009-08-12; First posted 2009-08-24 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-10

CONDITIONS: Blood Coagulation Disorders
Keywords: coumadine; genotype; genes; Warfarin
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinically Guided Cohort (Active Comparator): Estimated Effective Warfarin dosing calculations are based on clinical data algorithms
  Interventions: Drug: Warfarin
- Pharmacogenetically Guided Cohort (Experimental): Estimated Effective Warfarin dosing calculations are based on genetic and clinical data algorithms.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Dose estimates will be suggested daily for initial dose given and up to 4 consecutive doses after initial dose.
  Other Names: Coumadin

SUMMARY:
The purpose of this study is to explore how knowing genes that individuals inherit from their parents can make warfarin dosing more safe and effective. This study is being done to determine whether providing doctors with data on the genes their patients inherited and warfarin dosing recommendations based on those genes affects the costs and outcomes of care and after hospitalization for patients from different ethnic/racial backgrounds, and how physicians use this information in decision making.

DETAILED DESCRIPTION:
The overall goal of this project is to develop and assess the effectiveness and cost-effectiveness of strategies that use genetic testing in the management of anticoagulation among racially diverse hospitalized patients. The project has four specific aims.

Aim 1: To contribute patients initiating therapy at the University of Chicago Medical Center (UCMC) and affiliated hospitals to a genetic registry of a racially diverse set of patients undergoing warfarin therapy.

Aim 2: To perform a randomized trial to determine the efficacy, costs and cost-effectiveness of existing pharmacogenetic algorithms for the management of warfarin therapy among hospitalized patients of all races.

Aim 3: To develop clinical pharmacogenetic algorithms for the management of warfarin therapy among hospitalized African American patients.

Aim 4: To perform a randomized trial to determine and compare the efficacy, costs and cost-effectiveness of existing clinical and non-racially tailored pharmacogenetic algorithms to racially tailored pharmacogenetic algorithms for the management of warfarin therapy among hospitalized African American patients.

ELIGIBILITY:
Inclusion Criteria:

* warfarin-naive patients
* ages 18 and older
* are undergoing inpatient anticoagulation initiation with warfarin for diagnoses that necessitate anticoagulation

Exclusion Criteria:

* patients who are not warfarin-naive
* 17 years of age or younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O Meltzer, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were deleted from the study due to patient delay of surgery, baseline INR being too high, patient rescheduling or canceling surgery, no INR ordered, no admission to hospital.
Groups:
- Control: Control group received warfarin based on a clinically based dosing strategy during the first 6 days of therapy.
- Experimental: Experimental arm received warfarin based on a genotype based therapy during the first 6 days of therapy.
Period: Overall Study
Arm/Group | Control | Experimental
Started | 181 | 178
Completed | 181 | 178
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Estimated Effective Warfarin dosing calculations are based on clinical data algorithms
  Warfarin: Dose estimates will be suggested daily for initial dose given and up to 4 consecutive doses after initial dose.
- Experimental: Estimated Effective Warfarin dosing calculations are based on genetic and clinical data algorithms.
  Warfarin: Dose estimates will be suggested daily for initial dose given and up to 4 consecutive doses after initial dose.
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 181 | 178 | 359
Age, Customized [Count of Participants; unit: Participants] — Age categories are defined as 18-39, 40-60, 61-75, and 75 years and up.
  Participants
    18-39 years | 19 | 20 | 39
    40-60 years | 55 | 75 | 130
    61-75 years | 77 | 60 | 137
    75 years or more | 30 | 23 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 93 | 204
  Male | 70 | 85 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 171 | 170 | 341
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 84 | 72 | 156
  White | 85 | 93 | 178
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 181 | 178 | 359

OUTCOME MEASURES:

1. Primary Outcome: Inpatient Length of Stay
Description: Inpatient length of stay
Time Frame: during hospital stay, up to 60 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Experimental
Number analyzed (Participants) | 175 | 170
days | 6.8 (7.0) | 7.2 (11.2)

2. Secondary Outcome: Supratherapeutic Dosing
Description: International Normalized Ratio
Time Frame: during hospital stay, up to 60 days
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Control | Experimental
Number analyzed (Participants) | 175 | 170
ratio | 2.2 (0.2) | 2.2 (0.3)

ADVERSE EVENTS:
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/181 | 2/178
Serious Adverse Events (participants affected / at risk) | 7/181 | 1/178
Other Adverse Events (participants affected / at risk) | 0/181 | 0/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=181) | Experimental (N=178)
DVT or PE (Cardiac disorders) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No